CLINICAL TRIAL: NCT00273013
Title: Single Centre Allergen Challenge Study of GW274150 in Mild Asthmatic Subjects
Brief Title: Study With GW274150 In Patients With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: INO102141
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: asthma; allergen challenge
MeSH Terms: conditions — Asthma | interventions — GW 274150; montelukast

ARMS (6):
- Sequence 1 (Experimental): Subjects will receive Placebo in period 1, Singulair 10 milligrams (mg) in period 2 and GW274150 90 mg in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo
- Sequence 2 (Experimental): Subjects will receive Placebo in period 1, GW274150 90 mg in period 2 and Singulair 10 mg in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo
- Sequence 3 (Experimental): Subjects will receive Singulair 10 mg in period 1, Placebo in period 2 and GW274150 90 mg in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo
- Sequence 4 (Experimental): Subjects will receive Singulair 10 mg in period 1, GW274150 90 mg in period 2 and Placebo in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo
- Sequence 5 (Experimental): Subjects will receive GW274150 90 mg in period 1, Placebo in period 2 and Singulair 10 mg in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo
- Sequence 6 (Experimental): Subjects will receive GW274150 90 mg in period 1, Singulair 10 mg in period 2 and Placebo in period 3.
  Interventions: Drug: GW274150; Drug: Singulair; Drug: Placebo

INTERVENTIONS:
Drug: GW274150 — GW274150 will be available as 30 mg white oval tablets.
Drug: Singulair — Singulair will be available as over encapsulated 10 mg orange tablets.
  Other Names: GW274150
Drug: Placebo — Matching placebo for Singulair and GW274150 will be available.

SUMMARY:
This is a study investigating whether 14 days of dosing with GW274150 has a beneficial effect on a model of asthma type inflammation called the allergen-induced late asthmatic response. This will be compared with the response after treatment with a dummy (placebo) and a tablet treatment for asthma called Singulair (montelukast). Subjects in the study will receive all 3 treatments in a random order. The study is double-blind so subjects will not know which treatment they are taking at any given time.

ELIGIBILITY:
Inclusion criteria:

* Mild asthma: taking reliever medication (e.g. salbutamol) only.
* Screening involves measuring responses to the lung challenge agents: allergen, AMP, and methacholine. Only those with specific types of response to these will be eligible for the study.

Exclusion criteria:

* Recent steroid treatment.
* Significant illnesses or diseases other than asthma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-11-15 (Actual); Primary Completion 2005-10-28 (Actual); Study Completion 2005-10-28 (Actual)

PRIMARY OUTCOMES:
Effect on the late asthmatic reaction following an inhaled allergen challenge | Up to Day 115

SECONDARY OUTCOMES:
Measures of safety. Measures of lung function | Up to Day 115

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Singh D, Richards D, Knowles RG, Schwartz S, Woodcock A, Langley S, O'Connor BJ. Selective inducible nitric oxide synthase inhibition has no effect on allergen challenge in asthma. Am J Respir Crit Care Med. 2007 Nov 15;176(10):988-93. doi: 10.1164/rccm.200704-588OC. Epub 2007 Aug 23. PMID 17717202
- See also: Results for study 102141 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/INO102141?search=study&search_terms=102141#rs